CLINICAL TRIAL: NCT02149095
Title: A Phase I, Open-label, Dose Escalation Study to Determine the Maximum Tolerated Dose and Evaluate the Safety, Tolerability and Pharmacokinetics of Single Doses of TransCon PEG Treprostinil Administered as a Subcutaneous Injection in Healthy Adult Male Volunteers
Brief Title: Dose Escalation, MTD, Safety and PK Study of a Single Dose SC Injection of TransCon PEG Treprostinil in Healthy Male Volunteers
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study will not be conducted
Sponsor: United Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TCP-PH-101
Record Dates: First submitted 2014-05-20; First posted 2014-05-29 (Estimated); Last update posted 2014-08-07 (Estimated); Status verified 2014-08

CONDITIONS: PAH
Keywords: treprostinil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TransCon PEG treprostinil (Experimental): Dosing will begin at 0.116 mg/kg TransCon PEG treprostinil subcutaneous injection and the dose escalated in subsequent cohorts to MTD.
  Interventions: Drug: TransCon PEG treprostinil

INTERVENTIONS:
Drug: TransCon PEG treprostinil

SUMMARY:
TransCon PEG treprostinil is a novel prodrug form of treprostinil, in which treprostinil is reversibly conjugated via a four-arm branched polyethylene glycol (PEG) molecule. Reversible coupling of treprostinil to PEG should allow for a modified extended pharmacokinetic profile to achieve sustained plasma concentrations of treprostinil.

This will be the first investigation of TransCon PEG treprostinil in humans. This study aims to determine the maximum tolerated dose (MTD) and assess the safety, tolerability and pharmacokinetics of escalating single doses of a subcutaneous injection of TransCon PEG treprostinil.

ELIGIBILITY:
Inclusion Criteria:

1. Subject gives voluntary written informed consent to participate in the study
2. Subject is a healthy male between the ages of 18 and 50 years, inclusive, at Screening
3. Subjects must weigh between 60 and 120 kg, inclusive, with a BMI between 19.0-32.0 kg/m2, inclusive at Screening
4. Subject has a medical history, physical examination, vital signs, ECG and clinical laboratory results within normal limits or considered not clinically significant by the Investigator at Screening
5. Subject agrees to abstain from taking any prescription medication for 14 days prior to check-in and to abstain from taking any non-prescription medications (except multivitamins) or herbal supplements for 7 days prior to check-in Baseline until discharge from the study (unless prescribed by the Investigator to treat an AE)
6. Subject agrees to abstain from consuming alcohol from three days prior to check-in and until discharge from the study
7. Subject agrees to refrain from strenuous exercise from check-in and until discharge from the study
8. Subject is able to communicate effectively with study personnel and be considered reliable, willing and cooperative in terms of compliance with the protocol requirements

Exclusion Criteria:

1. Subject has any clinically relevant abnormality identified during the screening physical examination, 12-lead ECG, or laboratory examinations
2. Subject has a history of anaphylaxis, a previous documented hypersensitivity reaction, or a clinically significant idiosyncratic reaction to any drug
3. Subject has a clinically significant history of neurological, cardiovascular, respiratory, endocrine, hematological, hepatic, renal, gastrointestinal, genitourinary, pulmonary, and/or musculoskeletal disease; glaucoma; a psychiatric disorder, or any other chronic disease, whether controlled by medication or not
4. Subject has a history of postural hypotension, or unexplained syncope
5. Subject has a blood pressure that is less than 85 mmHg systolic or 50 mmHg diastolic at Screening or Baseline
6. Subject has a pulse rate that is greater than 90 bpm after sitting at rest for 5 minutes at Screening or Baseline
7. Subject has a history of hypertension
8. Subject has a blood pressure that is greater than 150 mmHg systolic or 90 mmHg diastolic at Screening or Baseline
9. Subject has a predisposing condition that could interfere with the absorption, distribution, metabolism, or excretion of drugs
10. Subject has tested positive at the screening visit for HIV infection, HBsAg, or the HCV antibody
11. Subject currently uses tobacco products or has a history of tobacco use within six months prior to Baseline
12. Subject has a history of alcohol abuse or a history of or current impairment of organ function reasonably related to alcohol abuse
13. Subject has a history of or current evidence of abuse of licit or illicit drugs or a positive urine screen for drugs of abuse
14. Subject has a history of abnormal bleeding tendencies
15. Subject has donated blood or plasma or has lost a significant volume of blood (greater than 450 mL) within four weeks prior to Baseline
16. Subject has participated in any investigational drug study within 30 days prior to Screening

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2014-07; Primary Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent AEs | Day 43
Maximum tolerated dose | 5 days
Treatment-emergent changes in clinical laboratory results | 43 days
Treatment-emergent changes in vital signs | 43 days

SECONDARY OUTCOMES:
Area under the concentration versus time curve: (AUC) | 42 days
Maximum observed plasma concentration: Cmax | 42 days
Time to maximum observed plasma concentration: Tmax | 42 days

CONTACTS AND LOCATIONS:
Locations (1):
- PPD Development, Austin, Texas, United States